CLINICAL TRIAL: NCT00299169
Title: Randomized Trial Comparing N of 1 Trials to Standard Practice to Improve Adherence to Statins in Patients With Diabetes
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: insufficient recruitment/enrollment
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-06-135; IRF-061-05
Record Dates: First submitted 2006-03-02; First posted 2006-03-06 (Estimated); Last update posted 2008-01-08 (Estimated); Status verified 2006-09

CONDITIONS: Diabetes; Cardiovascular Disease; Hyperlipidemia
Keywords: N of 1 trial; diabetes mellitus; HMG CoA Reductase Inhibitors; cardiovascular disease
MeSH Terms: conditions — Diabetes Mellitus; Cardiovascular Diseases; Hyperlipidemias | interventions — Single-Case Studies as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): N of 1 trials of statin therapy
  Interventions: Behavioral: N of 1 Trials
- 2 (Other): usual care
  Interventions: Behavioral: N of 1 Trials

INTERVENTIONS:
Behavioral: N of 1 Trials — N of 1 Trials of statin therapy
  Other Names: usual care

SUMMARY:
Patients who are intolerant of statins in routine practice, but who lack objective evidence of significant harm, will be randomized to receive statins by either n of 1 trials or standard practice. Our hypothesis is that n of 1 trials will improve statin adherence, thereby improving low density lipoprotein cholesterol (LDL-C) levels.

DETAILED DESCRIPTION:
Cholesterol lowering medications called "statins" decrease heart disease in people with diabetes but research shows that many patients are not taking these medications, sometimes because of side effects. In our experience, the side effects attributed to statin therapy are often subjective, non-specific, and not associated with objective evidence for a clinically important problem. The most common example is muscle cramps despite a normal CK level, but other symptoms include fatigue, GI intolerance, and neurological symptoms.

Traditionally, the effects of treatments are determined using randomized controlled trials. N of 1 trials minimize these biases through randomization, double-blinding, and multiple crossovers, and are therefore excellent tools to evaluate adverse effects of therapies when symptoms are non-specific and objective evidence for a causal relationship is ambiguous.

Patients who are intolerant of statins in routine practice, but who lack objective evidence of significant harm, will be randomized to receive statins by either n of 1 trials or standard practice. Our hypothesis is that n of 1 trials will improve statin adherence, thereby improving low density lipoprotein cholesterol (LDL-C) levels. Patients in the n of 1 trials group will be given 1 month courses of either simvastatin or placebo. Patients in the group who are receiving statins according to standard practice will be given a prescription by the doctor in the usual way.

At the end of the study, we will determine if more patients participating in n of 1 trials group are taking statins compared to the patients in the conventional group and if this leads to lower cholesterol levels. We plan to use the results of this small feasibility study to test the methods and to plan a larger study on the same question.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of type 1 or 2 diabetes
* Age 18-80 years
* Indication for a statin by the 2003 Canadian Diabetes Association (CDA) Clinical Practice Guidelines
* Willingness to re-try a statin despite previous apparent intolerance
* Provision of signed informed consent

Exclusion Criteria:

* Contraindication to a statin: previous rhabdomyolysis, active liver disease or unexplained persistent elevations of serum transaminases (CK, AST, ALT >three times upper limit of normal), pregnancy or lactation
* Impaired renal function: severe renal insufficiency (creatinine clearance <30 ml/min)
* Presence of a condition such as malignancy for which the one-year prognosis is poor
* Inability of the patient to comply with the rigorous conditions of the trial
* Any other condition deemed to render the study harmful to the participant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2006-09; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
mean LDL levels | end of study

SECONDARY OUTCOMES:
the proportions of participants taking statins at the end of the trial | end of study

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte G McDonald, MD, Principal Investigator — Western University, Canada
Locations (1):
- St. Joseph's Health Care London, London, Ontario, Canada